CLINICAL TRIAL: NCT05352022
Title: Lowering Food Insecurity and Improving Diabetes With Financial Incentives (LIFT-FINANCE)
Brief Title: Lowering Food Insecurity and Improving Diabetes With Financial Incentives
Acronym: LIFT-FINANCE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Rebekah Jo Walker, Associate Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PRO41475
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Monthly Unconditional Financial Incentive (Experimental): Individuals assigned to this group will receive diabetes education and a monthly incentive to supplement income and enhance ability to purchase healthy food options.
  Interventions: Behavioral: Monthly Unconditional Financial Incentive; Behavioral: Diabetes Education
- Monthly Unconditional Plus Healthy Food Purchasing Financial Incentive (Experimental): Individuals assigned to this group will receive diabetes education, a monthly incentive to supplement income and enhance ability to purchase healthy food options, and an additional weekly incentive if receipt for purchase of healthy food items from a grocery store is provided.
  Interventions: Behavioral: Monthly Unconditional Financial Incentive; Behavioral: Weekly Food Purchasing Financial Incentive; Behavioral: Diabetes Education
- Monthly Unconditional Plus Healthy Food Purchasing Plus Glycemic Control Financial Incentive (Experimental): Individuals assigned to this group will receive diabetes education, a monthly incentive to supplement income and enhance ability to purchase healthy food options, an additional weekly incentive if receipt for purchase of healthy food items from a grocery store is provided, and an incentive at the end of the study based on absolute drop in HbA1c.
  Interventions: Behavioral: Monthly Unconditional Financial Incentive; Behavioral: Weekly Food Purchasing Financial Incentive; Behavioral: Glycemic Control Financial Incentive; Behavioral: Diabetes Education

INTERVENTIONS:
Behavioral: Monthly Unconditional Financial Incentive — No requirements will be placed on how or where funds will be spent.
Behavioral: Weekly Food Purchasing Financial Incentive — Incentive for healthy food purchases
  Arms: Monthly Unconditional Plus Healthy Food Purchasing Financial Incentive; Monthly Unconditional Plus Healthy Food Purchasing Plus Glycemic Control Financial Incentive
Behavioral: Glycemic Control Financial Incentive — Incentive for absolute drop in HbA1c
  Arms: Monthly Unconditional Plus Healthy Food Purchasing Plus Glycemic Control Financial Incentive
Behavioral: Diabetes Education — mailed education information

SUMMARY:
The overarching aim of this proposal is to test the efficacy of financial incentives in improving HbA1c, blood pressure, and quality of life in food insecure adults with poorly controlled type 2 diabetes. Using a clinical trial design, the investigators will randomize food insecure adults with type 2 diabetes to one of three financial incentive structures in combination with monthly mailings that will include diabetes education, healthy recipes, and meal planning resources.

DETAILED DESCRIPTION:
Study Overview: The overarching aim of this proposal is to test the efficacy of financial incentives in improving HbA1c, blood pressure, and quality of life in food insecure adults with poorly controlled type 2 diabetes. Using a clinical trial design, the investigators will randomize 150 (50 per arm) food insecure adults with type 2 diabetes to one of three financial incentive structures in combination with monthly mailings that will include diabetes education, healthy recipes, and meal planning resources. Each individual will be followed for 6 months, with study visits at baseline, post-intervention (3-months), and 6 months. The primary outcome will be glycemic control (HbA1c) measured at 6 months post-randomization, while the secondary outcomes will include blood pressure and quality of life at 6 months post-randomization. Each outcome will be investigated for within group change and between group change. Finally, a cost and cost effectiveness analysis will be conducted to inform implementation in a broader population.

Patient Randomization. A permuted block randomization method will be used to assign subjects to control or intervention. The research assistant will collect eligibility information and enter it into the study database via the secured RedCap study website. Once eligibility is confirmed, the computer will generate the intervention assignment based on the pre-programmed randomization scheme. All subjects who are randomized will be entered into the study database and analyzed according to CONSORT guidelines .

Description of the LIFT-FINANCE Intervention. LIFT FINANCE is comprised of education and a structured financial incentive. All participants will receive a diabetes education booklet and monthly diabetes education modules mailed to their home, that will include healthy menu recommendations, meal planning resources, and healthy recipes that are affordable and easy to make. In addition, participants will receive one of three structured incentives:

Group 1: Monthly Unconditional Financial Incentive - this group will receive monthly unconditional incentive of $100 per month for 6 months to supplement income and enhance ability to purchase healthy food options. No requirements will be placed on how or where funds will be spent.

Group 2: Monthly Unconditional Plus Healthy Food Purchasing Financial Incentive - this group will receive monthly unconditional incentive of $100 per month for 6 months to supplement income and enhance ability to purchase healthy food options. In addition, participants will receive an additional $25 incentive per week if receipt for purchase of healthy food items from a grocery store is provided.

Group 3: Monthly Unconditional Plus Healthy Food Purchasing Plus Glycemic Control Financial Incentive - this group will receive monthly unconditional incentive of $100 per month for 6 months to supplement income and enhance ability to purchase healthy food options. In addition, participants will receive an additional $25 incentive per week if receipt for purchase of healthy food items from a grocery store is provided. Finally, participants will receive incentives for absolute drop in hemoglobin A1c at 6 months as follows: If HbA1c has dropped 2% or more from baseline, or absolute HbA1c is less than 7%, the additional incentive will be $150. If HbA1c has dropped between 1% to 1.9% from baseline the additional incentive will be $100. If HbA1c has dropped between 0.5% to 0.9% from baseline the additional incentive will be $50.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* clinical diagnosis of type 2 diabetes
* HbA1c of 9 or higher at screening visit
* screen positive for food insecurity using food insecurity risk tool
* ability to communicate in English

Exclusion Criteria:

* mental confusion on interview suggesting significant dementia
* participation in other diabetes clinical trial
* alcohol or drug abuse/dependency based on CAGE screening tool
* active psychosis or acute mental disorder
* life expectancy of less than 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic control (HbA1c) | 6-months post randomization
  Point of care A1c machine will be used to obtain HbA1c

SECONDARY OUTCOMES:
Blood pressure (both systolic and diastolic) | 6-months post randomization
  Blood pressure readings (both systolic and diastolic) will be obtained using automated BP monitors programmed to take 3 readings at 2 minute intervals and give average of the 3 readings
Quality of life as measured by the Short Form Health Survey (SF-12) | 6-months post randomization
  The Short Form Health Survey (SF-12) version 1, developed by Ware et al. in 1996 is a valid and reliable instrument that will be used to measure quality of life. Scores will be reported in physical health related (PCS) and mental health related (MCS). Scores range from 0 to 100 with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah J Walker, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker RJ, Knapp RG, Dismuke-Greer CE, Walker RE, Ozieh MN, Egede LE. Lowering the impact of food insecurity in African American adults with type 2 diabetes mellitus (LIFT-DM) - Study protocol for a randomized controlled trial. Contemp Clin Trials. 2020 Dec;99:106206. doi: 10.1016/j.cct.2020.106206. Epub 2020 Nov 7. PMID 33166622